CLINICAL TRIAL: NCT04608279
Title: Evolution of the Proteinuria / Creatininuria Ratio in the First Month of Life in the Preterm Infant
Brief Title: Urinary Creatinin/Protein Ratio in Preterms
Acronym: PROTI-PREMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/CHU/09
Record Dates: First submitted 2019-10-08; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Preterm Infant; Renal Failure
MeSH Terms: conditions — Premature Birth; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From the first days of life, the newborn presents a "physiological" proteinuria explained by the coexistence of a glomerular and tubular immaturity, all the more marked as the gestational age (GA) is weak. In the child term, proteinuria decreases the first month and its persistence is the marker of kidney damage. The persistence of proteinuria in preterm infants is also considered a marker of renal impairment; however, neither the "physiological" values nor the pattern of urinary excretion of proteins in the first month of life are known.

The proteinuria / creatininuria ratio is a validated indicator of proteinuria, as it is correlated with 24-hour urine proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Premature gestational age at birth superior or equal to 32 week of amenorrhea hospitalized in the intensive care unit or neonatal intensive care unit of the University Hospital of Reunion, southern site, Saint Pierre, in the first 24 hours of life
* Informed consent form Legal representant

Exclusion Criteria:

* Renal malformation known in antenatal

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature gestational age at birth superior or equal to 32 week of amenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Evolution in time of Ratio of proteinuria / creatininuria | Day 0, Day 2 or Day 3, Day 5 or Day 6, Week 2, Week 3, Week 4
  Ratio of proteinuria / creatinine to P1 (D0), P2 (D2 or D3), P3 (D5 or D6), P4 (W2), P5 (W3) and P6 (W4).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de La Réunion, Saint-Pierre, La Réunion, France

IPD SHARING:
Plan to Share IPD: No